CLINICAL TRIAL: NCT03143933
Title: Comparison Between IV Propofol and Propofol/ Fentanyl Anesthesia on Patients Surgical Stress Response Using BIS
Brief Title: Comparison Between IV Propofol and Propofol/ Fentanyl Anesthesia on Patients Stress Response
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, May Mohamed Abdalla, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PT (1490)
Record Dates: First submitted 2017-04-22; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Stress
Keywords: propofol, BIS, general anesthesia
MeSH Terms: interventions — Propofol; Fentanyl

ARMS (2):
- propofol (Active Comparator): this arm will receive propofol in induction of anesthesia and blood sample will be withdrawn before induction and another sample will be withdrawn after induction with 3 mins
  Interventions: Drug: Propofol
- propofol and fentanyl (Active Comparator): this arm will receive propofol and fentanyl in induction of anesthesia and blood sample will be withdrawn before induction and another sample will be withdrawn after induction with 3 mins
  Interventions: Drug: Propofol; Drug: Fentanyl

INTERVENTIONS:
Drug: Propofol — I.V propofol
Drug: Fentanyl
  Other Names: propofol
  Arms: propofol and fentanyl

SUMMARY:
It is hypothesized that propofol, when used in general anesthesia (GA) influence patient's stress status and consequently affect stress response parameters. Hence, the objective of the presented research is to assess whether the propofol has anti-stress effect or not in patients undergoing surgeries that require GA and classified as The American Society of Anesthesiologists physical status 1 (ASA PS1)

DETAILED DESCRIPTION:
* Forty patients will be divided into two groups of patients (n=20 each), where in the first group anesthesia induction will be with propofol as a single agent, while patients in the second group will be anesthetized by propofol/fentanyl and the depth of anesthesia will be determined by BIS score and will be kept at 40-60.
* In both groups, blood will be withdrawn to assess the possible effect of these medications on stress by measuring the following parameters:

I- Hemodynamic indicators II- Catecholamines . III- Fasting blood glucose IV- Insulin level V- Cortisol VI- Vasopressin

VII- Cytokines:

ELIGIBILITY:
Inclusion Criteria:

ASA1

Exclusion Criteria:

* Patients who refused to participate in the study or to sign the consent form
* The very young and very old patients
* Severely agitated (panicked).
* ASA1 patients who had bradycardia during propofol induction and was reversed with atropine.
* Patients with any of the following pathologies: liver, kidney, lung, or cardiac diseases, allergic to medicines, alcohol abuse, pregnant, or having endocrine or neuropsychiatric diseases. Moreover, those with sepsis syndrome with hemodynamic instability, hypothermia, and poorly controlled coagulopathy will not be enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Primary end point; assessment of change in blood biochemical indicators of surgical stress | blood sample will withdrawn before induction of anesthesia with 10 mins and after induction of anesthesia with 3 mins
  blood testing includes: Catecholamines 1. Epinephrine 2. Nor epinephrine
  , Fasting blood glucose, Insulin level, Cortisol, Vasopressin, and Cytokines

SECONDARY OUTCOMES:
Secondary end point; assessment of change in BIS number | BIS readings will be recorded before induction of anesthesia with 10 mins and after induction of anesthesia with 3 mins
Tertiary end point; assessment of change in blood pressure | blood pressure readings will be recorded before induction of anesthesia with 10 mins and after induction of anesthesia with 3 mins
Quaternary end point; assessment of change in heart rate | heart rate readings will be recorded before induction of anesthesia with 10 mins and after induction of anesthesia with 3 mins

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Aini, Cairo, Egypt